CLINICAL TRIAL: NCT01342770
Title: Pioglitazone as a Candidate Chemoprevention Agent for Lung Cancer: A Pilot Trial Using a Pre-surgical Model in Early Stage NSCLC
Brief Title: Pioglitazone Hydrochloride in Treating Patients With Stage IA-IIIA Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-03826; NCI-2011-03826 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MAYO-MAY10-15-02; N01-CN-2012-00042; CDR0000699459; MAY10-15-02 (Other: Mayo Clinic); MAY10-15-02 (Other: DCP); N01CN00042 (NIH); N01CN35000 (NIH); P30CA015083 (NIH)
Record Dates: First submitted 2011-04-23; First posted 2011-04-27 (Estimated); Results first posted 2015-10-06 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Stage IA Non-Small Cell Lung Carcinoma; Stage IB Non-Small Cell Lung Carcinoma; Stage IIA Non-Small Cell Lung Carcinoma; Stage IIB Non-Small Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pioglitazone hydrochloride) (Experimental): Patients receive pioglitazone hydrochloride PO QD for 14-42 days. Patients then undergo surgery.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Pioglitazone Hydrochloride; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pioglitazone Hydrochloride — Given PO
  Other Names: Actos; Pioglitazone.HCl
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot phase II trial studies how well pioglitazone works in treating patients with stage IA-IIIA non-small cell lung cancer. Pioglitazone hydrochloride may slow the growth of tumor cells and may be an effective treatment for non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the mechanism(s) of action of pioglitazone as a candidate chemopreventive agent for lung cancer by investigating the effects on Ki-67 defined in non-small cell lung cancer (NSCLC) tumor tissue.

SECONDARY OBJECTIVES:

I. To determine the effects of pioglitazone on multiple markers listed below:

* Tumor tissue: caspase-3, cyclin D1, p21/Waf1, peroxisome proliferative activated receptor, gamma (PPARγ), mucin 1 (MUC1).
* Premalignant tissue: Ki-67, caspase-3, PPARγ.
* Histologically normal tissue: Ki-67, PPARγ. II. To evaluate the toxicity and safety of pioglitazone in this patient population.

III. To analyze the expression of serum markers that are affected by pioglitazone.

IV. To describe the effects of limited treatment with pioglitazone on tumor metabolic activity as determined by FDG-PET (assessed before and after a minimum of 2 weeks of treatment).

OUTLINE:

Patients receive pioglitazone hydrochloride orally (PO) once daily (QD) for 14-42 days. Patients then undergo surgery.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or biopsy-proven NSCLC
* Willingness to provide biopsy tissue for correlative studies
* Candidate for pulmonary resection; must be able to schedule >= 14 days and =< 42 days between registration and surgery to allow for treatment with pioglitazone
* Ability to understand and the willingness to sign a written informed consent document
* Ability and willingness to swallow oral tablets
* Ability and willingness to undergo two bronchoscopies (before treatment and at the time of surgery)

  * For those participants who are undergoing mediastinoscopy as part of their standard-of-care, the pre-treatment bronchoscopy may be performed during the mediastinoscopy; if the participant remains eligible for definitive surgical resection after the mediastinoscopy, the participant may proceed to registration and pioglitazone treatment
* Current or former smoker with a >= 10 pack-year smoking history
* Women of child-bearing potential and men who agree to use adequate contraception for the duration of study participation; women must not be pregnant or lactating; women of child-bearing potential (women considered not of childbearing potential if they are at least two years postmenopausal and/or surgically sterile) must have used adequate contraception (abstinence; barrier methods such as intrauterine device [IUD], diaphragm with spermicidal gel, condom, or others; and hormonal methods such as birth control pills or others) since her last menses prior to study entry; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately

Exclusion Criteria:

* Receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pioglitazone
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating woman
* Currently treated diabetes
* Participants with >= class II New York Heart Association (NYHA) congestive heart failure or history of congestive heart failure
* Participants with >= grade 2 (moderate) edema
* Participants currently receiving an inhibitor of cytochrome P450 family 2, subfamily C, polypeptide 8 (CYP2C8) (gemfibrozil, ketoconazole, quercetin, trimethoprim), or an inducer of CYP2C8 (cortisol, dexamethasone, phenobarbital, rifampin), or cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) substrate
* Prior neoadjuvant therapy for NSCLC
* History of bladder cancer or in situ bladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Limburg, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten subjects were pre-registered at one Cancer Prevention Network (CPN) member organization from 2011 to 2013.
Pre-assignment Details: Four participants were deemed screen failures (3 without histologically-confirmed non-small cell lung cancer (NSCLC) and 1 with metastatic NSCLC and were excluded from all analyses.
Period: Overall Study
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who met eligibility criteria that were registered and received study agent.
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 64 [54 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 6
Baseline Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants]
  0=Asymptomatic and fully active | 5
  1=Symptomatic and fully ambulatory | 1
Smoking Status [Number; unit: participants]
  Former | 4
  Current | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Ki-67 by Immunohistochemistry (IHC)
Description: Changes in the expression levels of Ki-67 will be plotted graphically, and percent change in expression levels will be formally assessed using the paired t-test or the Wilcoxon signed rank test, if the assumptions of the t-test (i.e. normality) are not met.
Time Frame: Baseline and at the time of surgery, after 42 days of treatment
Population: Includes all registered participants with pre- and post-intervention tumor tissue samples except one participant who was deemed ineligible post-registration
Measure: Median (Full Range); unit: Percent change in Ki-67 measurements
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Number analyzed (Participants) | 5
Percent change in Ki-67 measurements | -20.0 [-40.0 to -11.1]
Statistical Analysis 1: Comparison: Treatment (Pioglitazone Hydrochloride); Test type: Superiority or Other; p = 0.06, Wilcoxon Signed Rank

2. Secondary Outcome: Change in Apoptosis Assessment (e.g., Caspase-3)
Description: Changes in the expression levels (or grades) from baseline (prior to intervention) to post-intervention (resected tumor sample) will be plotted graphically as well as formally assessed using the McNemar's tests (for categorical variables) or Wilcoxon signed rank tests (for continuous variables) respectively.
Time Frame: Baseline and at the time of surgery, after 42 days of treatment
Population: Data were not collected. Study team decision not to analyze this endpoint.
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Levels of Serum CA-153
Description: Each participant's pre- and post serum levels of CA-153 will be graphically represented and the mean levels analyzed using a paired t-test or Wilcoxon signed rank test, if the assumptions of the t-test are not met.
Time Frame: Baseline and at the time of surgery, after 42 days of treatment
Population: Data were not collected due to a study team decision not to analyze this endpoint.
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Levels of Serum CRP
Description: Each participant's pre- and post serum levels of CRP will be graphically represented and the mean levels analyzed using a paired t-test or Wilcoxon signed rank test, if the assumptions of the t-test are not met.
Time Frame: Baseline and at the time of surgery, after 42 days of treatment
Population: Data not collected due to a study team decision not to analyze this endpoint.
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Number analyzed (Participants) | 0

5. Secondary Outcome: Gene Expression Analysis of RNA From Bronchial Brush Cells
Description: For the gene expression profiles obtained from the data from normal bronchial brush cells, each participant's pre- and post gene expression will be graphically represented and the mean expression levels analyzed using a paired t-test or Wilcoxon signed rank test, if the assumptions of the t-test are not met.
Time Frame: Up to the time of surgery, after 42 days of treatment
Population: Data not collected due to a study team decision not to analyze this endpoint.
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Number analyzed (Participants) | 0

6. Secondary Outcome: Incidence of Adverse Events Graded According to Common Terminology Criteria for Adverse Events Version 4.0
Description: To evaluate the adverse events profile, the maximum grade for each type of adverse event will be recorded for each participant and frequency tables will be reviewed to determine the overall patterns. The number and severity of adverse events (both regardless of attribution as well as those that are at least possibly, probably, or definitely related) will be tabulated and summarized.
Time Frame: Up to the time of surgery, after 42 days of treatment
Population: Includes all registered eligible participants
Measure: Number; unit: participants
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Number analyzed (Participants) | 5
participants
  No Adverse Events | 3
  Grade 1 Adverse Events | 2

7. Secondary Outcome: Number of Participants With Clinical Response, Based on Response Evaluation Criteria in Solid Tumors ( RECIST) Version 1.1
Description: Clinical response rates will be summarized. Complete response (CR) is the disappearance of all non-nodal target lesions (TL) and each target lymph node (LN) must have reduction in short axis to <1.0cm. Partial Response (PR) is at least a 30% decrease in the sum of the longest diameters (LD) of the non-nodal TR and the short axis of the target LN with the baseline sum diameters (BSD) as reference. Progression (PD) is at least 1 new malignant lesion or LN whose short axis increased to >1.5 cm or at least a 20% increase in the sum of TL diameters with the minimum sum of diameters as reference.
Time Frame: Up to the time of surgery, after 42 days of treatment
Population: Data not collected due to a study team decision not to analyze this endpoint.
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With Complete Pathologic Response
Description: Complete pathologic response was defined as no viable residual tumor cells. Acellular residual mucin pools also considered a pathologic complete response.
Time Frame: Up to the time of surgery, after 42 days of treatment
Population: Includes all registered participants
Measure: Number; unit: participants
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Number analyzed (Participants) | 6
participants
  Complete Response | 1
  No Response | 5

9. Secondary Outcome: Percent Change in Cyclin D1
Description: Changes in the expression levels from baseline (prior to intervention) to post intervention (resected tumor sample) will be plotted graphically.
Time Frame: Baseline to the time of surgery, after 42 days of treatment
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent change in Cyclin D1 measurements
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Number analyzed (Participants) | 5
Percent change in Cyclin D1 measurements | -69 [-91 to 50]

10. Secondary Outcome: Percent Change in MUC1
Description: as for outcome 9
Time Frame: Baseline to the time of surgery, after 42 days of treatment
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent change in MUC1 measurements
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Number analyzed (Participants) | 5
Percent change in MUC1 measurements | 0 [-16.7 to 40]

11. Secondary Outcome: Percent Change in p21
Description: as for outcome 9
Time Frame: Baseline to the time of surgery, after 42 days of treatment
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent change in p21 measurements
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Number analyzed (Participants) | 5
Percent change in p21 measurements | -5 [-88.9 to 50]

12. Secondary Outcome: Percent Change in PPARy
Description: as for outcome 9
Time Frame: Baseline to the time of surgery, after 42 days of treatment
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent change in PPARy measurements
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Number analyzed (Participants) | 5
Percent change in PPARy measurements | 183.4 [0 to 1100]

13. Secondary Outcome: Percent Change in SUVmax From the PET Scan
Description: The percent change from pre to post-intervention in SUV max values will be summarized using descriptive statistics and simple graphical plots.
Time Frame: Baseline to the time of surgery, after 42 days of treatment
Population: Includes registered eligible participants with pre- and post-intervention PET/CT images obtained
Measure: Median (Full Range); unit: Percent change in tumor SUV max values
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Number analyzed (Participants) | 3
Percent change in tumor SUV max values | 0 [-15.4 to 0]

14. Secondary Outcome: Pre-intervention SUV of PET Scan
Description: The pre- and post-intervention SUV will be summarized using descriptive statistics and simple graphical plots.
Time Frame: Baseline
Population: Includes registered eligible participants with pre- and post-intervention PET/CT images obtained
Measure: Median (Full Range); unit: SUV
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Number analyzed (Participants) | 3
SUV | 13.0 [12.2 to 18.7]

15. Secondary Outcome: Post-intervention SUV of PET Scan
Description: The pre- and post-intervention SUV will be summarized using descriptive statistics and simple graphical plots.
Time Frame: Time of surgery, after 42 days of treatment
Population: Includes registered eligible participants with pre- and post-intervention PET/CT images obtained
Measure: Median (Full Range); unit: SUV
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Number analyzed (Participants) | 3
SUV | 12.2 [11.0 to 18.7]

ADVERSE EVENTS:
Arm/Group | Treatment (Pioglitazone Hydrochloride)
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pioglitazone Hydrochloride) (N=5)
Oral Pain (Gastrointestinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less